CLINICAL TRIAL: NCT04653376
Title: Possible Relationship Between Apoptosis and Endoplasmic Reticulum Stress in the Etiopathogenesis of Chronic Tonsillitis and Tonsillar Hypertrophy
Brief Title: Relationship of Endoplasmic Reticulum Stress and Tonsillar Tissue Diseases
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merih Onal, Assistant Professor, Selcuk University
Other Study IDs: 2018/329
Record Dates: First submitted 2020-11-05; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Tonsillitis; Tonsillar Hypertrophy; Immune System Diseases
Keywords: Endoplasmic Reticulum; Apoptosis; İmmune system
MeSH Terms: conditions — Tonsillitis; Immune System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tonsillar tissues were gathered in groups in accordance with their size and analyzed in regards to Endoplasmic Reticulum stress and apoptosis markers by Real-Time PCR and Western Blotting method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic tonsillitis: Patients with tonsil sizes grade 1 and 2, and tonsillectomy indications included frequently recurrent tonsillary infection, sore throat, and malodorous mouth problems were accepted as the chronic tonsillitis group.
  Interventions: Procedure: Tonsillectomy surgery
- Tonsillar hypertrophy: Patients with tonsil size grades 3 and 4 and tonsillectomy indications included obstructive symptoms such as snoring, open mouth breathing, difficulty in breathing, and swallowing problems were accepted as the tonsillar hypertrophy group.
  Interventions: Procedure: Tonsillectomy surgery

INTERVENTIONS:
Procedure: Tonsillectomy surgery — The tonsillectomy procedure was performed under general anesthesia using the classical dissection method. Extracted tonsil tissue samples were sent to the medical genetics department in tubes to investigate the ER stress and apoptosis.

SUMMARY:
Tonsillar tissue is a significant organ for the performing of immune systems in children. The Endoplasmic Reticulum (ER), is an organelle needed for the care of a stable function of the cells. The purpose of the study was to explore the correlation among ER stress and tonsillar tissue disorders and to explain the structure of diseases related to the immune system.

DETAILED DESCRIPTION:
A prospective study was conducted on 46 children aged who underwent tonsillectomy for chronic tonsillitis or tonsil hypertrophy. Tonsil tissues were evaluated in terms of ER stress markers and apoptosis markers by Real-time PCR and Western blot methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent tonsillectomy surgery with the clinical diagnosis of chronic tonsillitis and tonsillar hypertrophy.

Exclusion Criteria:

* Systemic diseases
* Other otolaryngological disorders

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who underwent tonsillectomy surgery aged between 2 and 16 years and who were clinically diagnosed with chronic tonsillitis and tonsil hypertrophy by the ENT clinician.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Relationship of Endoplasmic Reticulum stress and apoptosis with chronic tonsillitis and tonsillar hypertrophy | 2018-2020
  Our primary outcome was to evaluate providing that Endoplasmic Reticulum stress and apoptosis reaction performing in chronic tonsillitis and tonsillar hypertropy, which is related with the immune system of children. GRP78, CHOP, ATF6, ATF4 proteins will be investigated in tonsillar tissues to evaluate ER stress index, and bax, bcl2 proteins will be investigated to evaluate apoptosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We will share the study protocol after our article has been accepted for publication in a journal.

REFERENCES:
- [Background] So JS. Roles of Endoplasmic Reticulum Stress in Immune Responses. Mol Cells. 2018 Aug 31;41(8):705-716. doi: 10.14348/molcells.2018.0241. Epub 2018 Jul 30. PMID 30078231
- [Background] Onal M, Yilmaz T, Bilgic E, Muftuoglu SF, Kuscu O, Gunaydin RO. Apoptosis in chronic tonsillitis and tonsillar hypertrophy. Int J Pediatr Otorhinolaryngol. 2015 Feb;79(2):191-5. doi: 10.1016/j.ijporl.2014.12.005. Epub 2014 Dec 15. PMID 25555639
- [Derived] Onal M, Kocak N, Duymus F, Bozkurt MK, Elsurer C, Erdur O, Onal O. Relationship of endoplasmic reticulum stress with the etiopathogenesis of chronic tonsillitis and tonsillar hypertrophy in pediatric patients: a prospective, parallel-group study. Mol Biol Rep. 2021 Jul;48(7):5579-5586. doi: 10.1007/s11033-021-06579-4. Epub 2021 Jul 22. PMID 34292473